CLINICAL TRIAL: NCT01748058
Title: Active Video Games to Promote Physical Activity, Motor Performance and Quality of Life in Children With Cancer: an Intervention Study With 2-year Follow-up
Brief Title: Active Video Games to Promote Physical Activity in Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Päivi Lähteenmäki, MD, PhD, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: T87/2012
Record Dates: First submitted 2012-10-15; First posted 2012-12-12 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

ARMS (2):
- Active video games (Experimental): Exercise based on active video gaming
  Interventions: Behavioral: Exercise based on active video gaming
- Routine care (No Intervention)

INTERVENTIONS:
Behavioral: Exercise based on active video gaming
  Arms: Active video games

SUMMARY:
The aim of this study is to evaluate the efficacy and feasibility of active video gaming with regard to the promotion of physical activity and motor learning in children with cancer. Experienced fatigue, body mass index and the development of metabolic risk factors during treatment are also examined.

ELIGIBILITY:
Inclusion Criteria:

* cancer diagnose
* treated with Vincristine in Turku University Hospital or Tampere University Hospital

Exclusion Criteria:

* other diseases limiting functional ability
* not able to communicate

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Accelerometer, average counts of dynamic acceleration (physical activity) | 1 week at baseline and at 12 months
  Change in the children's physical activity levels with accelerometer

SECONDARY OUTCOMES:
Movement assessment battery for children (M-ABC-2) scores (motor performance) | At baseline, 2, 6, 12 and 24 months
  Change in M-ABC scores
PedsQL Multidimensional Fatigue Scale scores (fatigue) | At baseline, 2, 6, 12 and 24 months
  Change in experienced fatigue
Blood sugar | At baseline, 2, 6, 12 and 24 months
  Change in blood sugar
Blood insulin | At baseline, 2, 6, 12 and 24 months
  Change in blood insulin

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Hamari L, Jarvela LS, Lahteenmaki PM, Arola M, Axelin A, Vahlberg T, Salantera S. The effect of an active video game intervention on physical activity, motor performance, and fatigue in children with cancer: a randomized controlled trial. BMC Res Notes. 2019 Nov 29;12(1):784. doi: 10.1186/s13104-019-4821-z. PMID 31783907
- [Derived] Kauhanen L, Jarvela L, Lahteenmaki PM, Arola M, Heinonen OJ, Axelin A, Lilius J, Vahlberg T, Salantera S. Active video games to promote physical activity in children with cancer: a randomized clinical trial with follow-up. BMC Pediatr. 2014 Apr 5;14:94. doi: 10.1186/1471-2431-14-94. PMID 24708773
- See also: Study protocol — http://www.biomedcentral.com/1471-2431/14/94
- See also: Results — https://bmcresnotes.biomedcentral.com/articles/10.1186/s13104-019-4821-z